CLINICAL TRIAL: NCT06722209
Title: Investigation of the Effect of Different Same-day Colonoscopic Bowel Preparation Procedures on Patient Compliance, Tolerability, and Bowel Cleansing: a Randomized Controlled Trial
Brief Title: Different Same-day Colonoscopic Bowel Preparation Procedures on Patient Compliance, Tolerability, and Bowel Cleansing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülten Sucu Dağ, Assoc Prof, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GSD-3
Record Dates: First submitted 2024-11-29; First posted 2024-12-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Colonoscopy; Colonoscopy Diagnostic Techniques and Procedures; Colonoscopy Preparation; Colonoscopy Preparation Outcome
Keywords: Colonoscopy; Bowel preparation; Colorectal cancer; Patients compliance
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial with experimental and control groups
Who Masked: Outcomes Assessor
Masking Description: The statistician will not know which group the intervention is for. Data entry will be made as A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Intervention group (Other): Intestinal preparation protocol with polyethylene glycol (Protocol I)
  Interventions: Other: polyethylene glycol (Protocol I)
- Control group (Other): Intestinal preparation protocol with with sodium phosphate content (protocol II)
  Interventions: Other: polyethylene glycol (Protocol I)

INTERVENTIONS:
Other: polyethylene glycol (Protocol I) — Intestinal preparation protocol with polyethylene glycol (Protocol I)

SUMMARY:
The aim of this study was to investigate the effect of different bowel preparation protocols applied on the same day on patients' compliance, tolerance and bowel cleansing before colonoscopy.

Hypotheses of the Study : Same-day administration of bowel preparation before colonoscopy; H1.1: There is a significant difference between the bowel preparation protocol with polyethylene glycol (Protocol I) and the protocol with sodium phosphate (Protocol II) in bowel preparation score scores H1.2: There is a significant difference between the compliance levels of the patients who underwent a bowel preparation protocol containing polyethylene glycol (Protocol I) and a protocol containing sodium phosphate (Protocol II) H1.3: There is a significant difference between the tolerance of the patients who underwent a bowel preparation protocol containing polyethylene glycol (Protocol I) and a protocol containing sodium phosphate (Protocol II)

In patients in Protocol I and II groups, data will be collected one day before the procedure with the Descriptive Characteristics Form and the procedure will be explained face to face. After the procedure, bowel preparation score during colonoscopy and compliance and tolerance to the bowel preparation protocol will be evaluated from the patients in both groups.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of different bowel preparation protocols applied on the same day on patients' compliance, tolerance and bowel cleansing before colonoscopy.

This study will be conducted as a single centre prospective randomised controlled trial in accordance with the principles of the Declaration of Helsinki. The study will be conducted in a private clinic in Famagusta region in patients undergoing colonoscopy.

Patients undergoing colonoscopy will be given written material about bowel preparation the day before the procedure and the protocol will be explained verbally and in writing. The bowel preparation protocol is described below.

Protocol I 06.30 Breakfast 09.00 hours: Phospho-Soda 45 ml 10.00: Phospho-Soda 45 ml At least 3 litres of liguid fluid intake until 14.00 14.30- 15.00: Colonoscopy Protocol II 06.30 Breakfast 09.00 :Polyethylene Glycol (PEG) will be diluted with 4 litres of water and one glass (200ml) will be drunk every 10 minutes until it is finished (It will be finished in about 4 hours) Colonoscopy after 2 hours Inclusion criteria

* Over 18 years of age
* Drinking at least 75 per cent of the solution
* Have the ability to read and understand research instructions
* Patients who agreed to participate in the study Sampling exclusion criteria
* Patients with active lower intestinal bleeding Patients diagnosed with CHF, liver failure, end-stage acute renal failure

A total of 118 patients were planned to be included in the study with an effect size of d=0.50, α =0.05 margin of error, 85% power, and 59 patients in each group. Considering the possibility of missing data, the sample number was increased by 10% and it was decided to take 128 patients by taking 64 patients in the groups in total.

The patients will be assigned to the experimental and control groups according to the list to be created using the randomisation program at a ratio of 1.1(https://www.random.org/). Randomisation and assignment to groups will be done by an independent researcher who is not involved in the implementation phase of the research. Thus, selection bias will be prevented in the randomization process.

In patients in Protocol I and II groups, data will be collected one day before the procedure with the Descriptive Characteristics Form and the procedure will be explained face to face. After the procedure, the bowel preparation score during colonoscopy and compliance and tolerance to the bowel preparation protocol will be evaluated from the patients in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Drinking at least 75 per cent of the solution
* Have the ability to read and understand research instructions
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients with active lower intestinal bleeding
* KKY
* Liver failure,
* Patients with end-stage acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Compliance and Tolerance to the Bowel Preparation Protocol | The patients were interviewed 30-60 dk minutes after the procedure was completed.
  The Bowel Preparation Protocol Compliance and Tolerance Assessment Form will assess this primary outcome. This form assesses tolerance to the bowel preparation protocol; abdominal pain, nausea, vomiting, Abdominal distension -gas,thirst , headache, weakness and fatigue and intolerance to the solution. The rate of patients experiencing variables including Compliance and Tolerance to the Bowel Preparation Protocol will be calculated.

SECONDARY OUTCOMES:
Bowel cleansing quality level | BBPS will be assessed by the surgeon during colonoscopy.
  The effect of the bowel preparation protocol on bowel readiness will be assessed using the Boston Bowel Readiness Classification. Boston Classification of Bowel Preparation (BBPS) scores bowel cleanliness between 0 and 3 points. According to BBPS, 3 segments of the colon (left, transverse, right) are scored according to the degree of cleanliness. According to BBPS, a score of 0 indicates inadequate cleanliness and a score of 9 indicates perfect cleanliness. As the cleanliness score progresses from zero to nine, it is assessed that bowel cleanliness is approaching perfection.

REFERENCES:
- [Background] Theunissen F, Lantinga MA, Ter Borg PCJ, Ouwendijk RJT, Siersema PD, Bruno MJ; Trans. IT foundation study group. Efficacy of different bowel preparation regimen volumes for colorectal cancer screening and compliance with European Society of Gastrointestinal Endoscopy performance measures. United European Gastroenterol J. 2023 Jun;11(5):448-457. doi: 10.1002/ueg2.12386. Epub 2023 May 15. PMID 37190897
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37190897/